CLINICAL TRIAL: NCT03781375
Title: A Phase III Double Blind Randomized Study Comparing Etanercept (Enbrel) Combined With Methotrexate vs Methotrexate Alone in Children With Polyarticular Course Juvenile Rheumatoid Arthritis
Brief Title: Etanercept Plus Methotrexate Versus Methotrexate Alone in Children With Polyarticular Course Juvenile Rheumatoid Arthritis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20021628; 016.0028 (Other: Immunex Corporation)
Record Dates: First submitted 2018-12-18; First posted 2018-12-19 (Actual); Results first posted 2019-08-02 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-06

CONDITIONS: Juvenile Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Juvenile | interventions — Etanercept; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Methotrexate + Placebo (Placebo Comparator): Participants received placebo subcutaneous injections twice weekly and methotrexate once a week at the same dose as prior to study entry for 6 months. After month 6 participants received open-label 0.4 mg/kg etanercept twice weekly plus methotrexate for an additional 6 months.
  Interventions: Drug: Etanercept; Drug: Placebo to Etanerceot; Drug: Methotrexate
- Methotrexate + Etanercept (Experimental): Participants received 0.4 mg/kg etanercept subcutaneous injections twice weekly and methotrexate once a week at the same dose as prior to study entry for 6 months. After month 6 participants received open-label 0.4 mg/kg etanercept twice weekly plus methotrexate for an additional 6 months.
  Interventions: Drug: Etanercept; Drug: Methotrexate

INTERVENTIONS:
Drug: Etanercept — Administered by subcutaneous injection twice a week
  Other Names: Enbrel
Drug: Placebo to Etanerceot — Administered by subcutaneous injection twice a week
  Arms: Methotrexate + Placebo
Drug: Methotrexate — Administered orally or subcutaneously once a week at the same dose as prior to study entry

SUMMARY:
The primary objective of this study was to determine the efficacy of etanercept plus methotrexate vs methotrexate alone in pediatric patients with active polyarticular course juvenile rheumatoid arthritis (JRA).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have had a diagnosis of JRA by the American College of Rheumatology (ACR) criteria. Disease onset may have been systemic, polyarticular, or pauciarticular
* Disease course must have been polyarticular with at least 5 active joints
* Duration of disease was not limited, but must have been long enough for the patient to have been given a 3-month trial of non-steroidal anti-inflammatory drugs (NSAIDs) and methotrexate at a dose between 0.3 and 1.0 mg/kg/week, orally (PO) or subcutaneously (SC)
* Receiving methotrexate at a dose between 0.3 mg/kg/wk and 1 mg/kg/wk at time of randomization. The dose of methotrexate must have been stable for one month prior to entry
* Patients may have failed prednisone, or been on a dosage of prednisone not to have exceeded 10 mg/day or 0.20 mg/kg/day (whichever was less)
* At the time of qualification (screening) for study and prior to wash-out of all disease modifying anti-rheumatic drugs (DMARDs), the patient must have had active disease, defined as ≥ 5 swollen joints accompanied by pain, and/or tenderness and/or warmth, and ≥ 3 joints with limitation of motion (LOM). (The joints with LOM may have been the same as those with swelling)
* Had good venous access and stable hematocrit ≥ 24 mL/dL
* Patients must have been pre-pubescent, or if post-pubertal at anytime during the study, and of child-bearing potential, must have been practicing adequate contraception
* Parent or legal guardian was able and willing to give informed consent
* Parent or legal guardian must have been willing to actively supervise storage and administration of study drug and ensure that the date and time of each dose was accurately recorded in the subject's diary

Exclusion Criteria:

* Was unable to meet the concurrent medication restrictions as described in the protocol
* Pregnant or nursing female
* Patients were excluded if they demonstrated clinically significant deviations from normal (as defined below) in any of the following laboratory parameters:

  * thrombocytopenia; platelet count < 100,000/cmm
  * leukopenia; total white cell count < 4000 cells/cmm
  * neutropenia; neutrophils < 1000 cells/cmm
  * hepatic transaminase levels > two times the upper limit of normal (ULN)
  * serum bilirubin > two times the ULN
  * estimated creatinine clearance of < 90 mL/min/1.73 M² body surface area (BSA)
  * known human immunodeficiency virus (HIV), hepatitis B surface antigen positivity not related to vaccination, or hepatitis C antibody positivity
* Had received etanercept, antibody to tumor necrosis factor (TNF) (i.e. infliximab or D2E7), antibody to cluster of differentiation (CD)4 (anti-CD4), diphtheria interleukin (IL)-2 fusion protein (DAB-IL-2) or leflunomide
* Had received DMARDs including D-penicillamine, hydroxychloroquine, sulfasalazine, oral or injectable gold, cyclosporin, azathioprine; intravenous immunoglobulin (IV Ig); or broadly immunosuppressant chemotherapeutic agents (e.g. cyclophosphamide, FK506, mycophenolate mofetil [CellCept]), for at least 28 days prior to enrollment and dosing of study drug. All DMARDs, other than methotrexate, must have been washed-out for a minimum of 28 days
* Had received intraarticular glucocorticoid injection within 28 days prior to enrollment on study
* Had previously received live virus vaccine within 3 months prior to study entry
* Had participated in a study of an investigational drug or biologic requiring informed-consent within three months prior to study entry
* Any concurrent medical condition which would have, in the investigator's opinion, compromised the patient's ability to tolerate the study drug or would have made the patient unable to cooperate with the protocol
* History of/or current psychiatric illness that would have interfered with ability to comply with protocol requirements or give informed consent
* Chronic or recurrent infections, or currently active infection at screening
* History of alcohol or drug abuse that would have interfered with ability to comply with protocol requirements
* Inability to have complied with the study requirements

Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2000-08-24 (Actual); Primary Completion 2002-06-20 (Actual); Study Completion 2002-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 7 centers in the United States. The study consisted of a 6-month double-blind treatment period followed by a 6-month open-label period where all participants received etanercept + methotrexate. Early transition to open-label treatment was allowed after 2 months of blinded treatment, for disease flare or lack of response.
Pre-assignment Details: Participants were randomized equally into 1 of 2 treatments for the double-blind portion of the study. Randomization was stratified by route of methotrexate administration (oral [PO] vs subcutaneous [SC]) prior to randomization.
Period: Double-blind Phase
Arm/Group | Methotrexate + Placebo | Methotrexate + Etanercept
Started | 12 | 13
Received Study Drug | 12 | 13
Completed | 5 | 7
Not Completed | 7 | 6
Not completed — Adverse Event | 0 | 1
Not completed — Lack of Response | 6 | 2
Not completed — Other | 1 | 3
Period: Open-label Phase
Arm/Group | Methotrexate + Placebo | Methotrexate + Etanercept
Started (Participants who completed blinded treatment or who withdrew early due to flare or lack of response) | 11 | 9
Received Study Drug | 10 | 9
Completed | 8 | 6
Not Completed | 3 | 3
Not completed — Protocol Issues | 0 | 1
Not completed — Suboptimal Clinical Response | 1 | 0
Not completed — Other | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Methotrexate + Placebo | Methotrexate + Etanercept | Total
Number analyzed (Participants) | 12 | 13 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.75 (5.71) | 11.38 (3.40) | 10.12 (4.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 5 | 7 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 10 | 10 | 20
  Black | 2 | 0 | 2
  Hispanic | 0 | 2 | 2
  Oher | 0 | 1 | 1
Methotrexate Dosage Route [Count of Participants; unit: Participants] — Randomization was stratified on methotrexate dose route.
  Participants
    Orally | 5 | 6 | 11
    Subcutaneously | 7 | 7 | 14
Type of Arthritis at Onset [Count of Participants; unit: Participants]
  Pauciarticular | 1 | 4 | 5
  Polyarticular | 7 | 9 | 16
  Systemic | 4 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a JRA Response at Month 6
Description: Response was defined using the JRA definition of improvement (JRA DOI) as a ≥ 30% improvement from baseline in at least three of the six JRA Core Set Criteria and ≥ 30% worsening in not more than one of the six assessments. The JRA Core Set Criteria consist of:
  * Physician's global assessment of disease severity assessed on a visual analog scale (VAS) from 1 to 10
  * Patient's/Parent's global assessment of overall well being assessed on a VAS from 1 to 10
  * Number of active joints (swelling, not due to deformity, or if no swelling is present, limitation of motion accompanied by pain on passive motion and/or tenderness and/or warmth)
  * Number of joints with limitation of motion
  * Childhood Health Assessment Questionnaire (CHAQ)
  * Erythrocyte sedimentation rate (ESR)
Time Frame: Baseline and month 6
Population: All randomized participants; participants with missing data are counted as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Methotrexate + Placebo | Methotrexate + Etanercept
Number analyzed (Participants) | 12 | 13
percentage of participants | 33 | 38

2. Secondary Outcome: Percentage of Participants With a 50% Improvement in JRA DOI at Month 6
Description: Response was defined using the JRA definition of improvement (JRA DOI) as a ≥ 50% improvement from baseline in at least three of the six JRA Core Set Criteria and ≥ 30% worsening in not more than one of the six assessments. The JRA Core Set Criteria consist of:
  * Physician's global assessment of disease severity assessed on a visual analog scale (VAS) from 1 to 10
  * Patient's/Parent's global assessment of overall well being assessed on a VAS from 1 to 10
  * Number of active joints (swelling, not due to deformity, or if no swelling is present, limitation of motion accompanied by pain on passive motion and/or tenderness and/or warmth)
  * Number of joints with limitation of motion
  * Childhood Health Assessment Questionnaire (CHAQ)
  * Erythrocyte sedimentation rate (ESR)
Time Frame: Baseline and month 6
Population: All randomized participants; participants with missing data were counted as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Methotrexate + Placebo | Methotrexate + Etanercept
Number analyzed (Participants) | 12 | 13
percentage of participants | 25 | 38

3. Secondary Outcome: Percentage of Participants With a 70% Improvement in JRA DOI at Month 6
Description: Response was defined using the JRA definition of improvement (JRA DOI) as a ≥ 70% improvement from baseline in at least three of the six JRA Core Set Criteria and ≥ 30% worsening in not more than one of the six assessments. The JRA Core Set Criteria consist of:
  * Physician's global assessment of disease severity assessed on a visual analog scale (VAS) from 1 to 10
  * Patient's/Parent's global assessment of overall well being assessed on a VAS from 1 to 10
  * Number of active joints (swelling, not due to deformity, or if no swelling is present, limitation of motion accompanied by pain on passive motion and/or tenderness and/or warmth)
  * Number of joints with limitation of motion
  * Childhood Health Assessment Questionnaire (CHAQ)
  * Erythrocyte sedimentation rate (ESR)
Time Frame: Baseline and month 6
Population: All randomized participants; participants with missing data were counted as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Methotrexate + Placebo | Methotrexate + Etanercept
Number analyzed (Participants) | 12 | 13
percentage of participants | 8 | 38

ADVERSE EVENTS:
Time Frame: Up to 12 months on-study evaluations plus 1 month follow-up
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Groups:
- Methotrexate + Placebo (Blinded Phase): Participants received placebo subcutaneous injections twice weekly and methotrexate once a week at the same dose as prior to study entry for 6 months.
- Methotrexate + Etanercept (Blinded Phase): Participants received 0.4 mg/kg etanercept subcutaneous injections twice weekly and methotrexate once a week at the same dose as prior to study entry for 6 months.
- Methotrexate + Etanercept (Open Label Phase): After month 6 participants received open-label 0.4 mg/kg etanercept twice weekly plus methotrexate for an additional 6 months.
Arm/Group | Methotrexate + Placebo (Blinded Phase) | Methotrexate + Etanercept (Blinded Phase) | Methotrexate + Etanercept (Open Label Phase)
Serious Adverse Events (participants affected / at risk) | 1/12 | 1/13 | 0/19
Other Adverse Events (participants affected / at risk) | 11/12 | 12/13 | 15/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Methotrexate + Placebo (Blinded Phase) (N=12) | Methotrexate + Etanercept (Blinded Phase) (N=13) | Methotrexate + Etanercept (Open Label Phase) (N=19)
Appendicitis (Infections and infestations) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Methotrexate + Placebo (Blinded Phase) (N=12) | Methotrexate + Etanercept (Blinded Phase) (N=13) | Methotrexate + Etanercept (Open Label Phase) (N=19)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 2 | 1
Cerumen impaction (Ear and labyrinth disorders) | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0
Blepharospasm (Eye disorders) | 1 | 0 | 0
Uveitis (Eye disorders) | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 3 | 2
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1 | 2
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 0 | 3
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 3 | 3
Chest pain (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0
Injection site erythema (General disorders) | 0 | 1 | 0
Injection site pain (General disorders) | 0 | 1 | 0
Injection site pruritus (General disorders) | 0 | 0 | 1
Injection site rash (General disorders) | 0 | 1 | 1
Injection site reaction (General disorders) | 0 | 0 | 3
Oedema peripheral (General disorders) | 0 | 0 | 1
Pain (General disorders) | 0 | 1 | 1
Peripheral swelling (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 2 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 1
Beta haemolytic streptococcal infection (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0
Chronic sinusitis (Infections and infestations) | 0 | 1 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 2
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
Otitis media (Infections and infestations) | 2 | 0 | 3
Pharyngitis (Infections and infestations) | 0 | 1 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 2
Sinusitis (Infections and infestations) | 2 | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 2 | 4 | 2
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Mouth injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1
Blood pressure diastolic increased (Investigations) | 0 | 1 | 0
Body temperature increased (Investigations) | 1 | 0 | 1
Liver function test increased (Investigations) | 1 | 0 | 0
Lymph node palpable (Investigations) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 3 | 6 | 3
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0
Tongue biting (Nervous system disorders) | 0 | 0 | 1
Aggression (Psychiatric disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1
Tic (Psychiatric disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 3
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pseudoporphyria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 3 | 4
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin atrophy (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin burning sensation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hot flush (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.